CLINICAL TRIAL: NCT00669110
Title: 6-Month, Multicenter, Open-Label, Flexible-Dose Study To Evaluate Safety, Efficacy, And Tolerability Of Desvenlafaxine Succinate Sustained-Release Tablets In The Treatment Of Child And Adolescent Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained-Release Tablets (DVS SR) In The Treatment Of Child and Adolescent Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A6-2001; B2061013
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Depressive Disorder, Major Depressive Disorder
Keywords: MDD; Depression; Pediatrics; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Tablets (DVS SR)

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release Tablets (DVS SR) — * tablet
  * subjects randomly assigned to 10-200 mg/day by age group
  * 6 month treatment period(~182 days)

SUMMARY:
The primary purpose of this study is to evaluate the long-term safety and tolerability of Desvenlafaxine Succinate Sustained-Release (DVS SR) in child and adolescent outpatients with major depressive disorder. A secondary aim is to evaluate the efficacy of DVS SR in the treatment of child and adolescent outpatients with major depressive disorder in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed 8-weeks of treatment in the preceding study, 3151A6-2000, and who, in the opinion of the investigator, would benefit from long-term treatment.
* Study participants who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 15 days after the last dose of test article. Sexually active study participants must agree and commit to the use of condoms in addition to other contraceptive methods.

Exclusion Criteria:

* Clinically important abnormalities on baseline physical examination or any clinically significant abnormality on electrocardiogram (ECG), laboratory test results, or vital signs recorded before the final study day (day 56 visit) of the preceding study 3151A6-2000.
* Unresolved clinically significant adverse events or serious adverse events in the preceding study 3151A6-2000.
* Poor compliance with the preceding study 3151A6-2000, as assessed by the investigator and the medical monitor.
* Other exclusion criteria apply.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (9):
- United States (9):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A6-2001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants transitioned from preceding Core study NCT00619619 (3151A6-2000 [B2061012]) on Day 56 to this Extension study NCT00669110 (3151A6-2001 [B2061013]) to continue treatment on a flexible dose schedule. A total of 8 participants (Children n=2 and Adolescent n=6) discontinued during Taper/post-study or Follow-up phase of Core study.
Pre-assignment Details: Baseline (Day-1) in the Extension study = Week 8 (Day 56) in the Core study. However, Baseline for the Clinical Global Impressions Scale - Improvement (CGI-I) = Inpatient Day 1 through 4 in the Core study and Baseline for the Columbia Suicide-Severity Rating Scale (C-SSRS) = Day-1 in the Core study.
Groups:
- DVS SR - Children: Desvenlafaxine succinate sustained-release (DVS SR) formulation tablet(s) by mouth (PO) administered as flexible dosing adjusted by the investigator as clinically indicated. Total daily dose will be flexible between 10 milligrams (mg), 25 mg, 50 mg, and 100 mg for children 7 to 11 years of age at baseline in the preceding Core study NCT00619619.
- DVS SR - Adolescents: Desvenlafaxine succinate sustained-release (DVS SR) formulation tablet(s) by mouth (PO) administered as flexible dosing adjusted by the investigator as clinically indicated. Total daily dose will be flexible between 25 mg, 50 mg, 100 mg, and 200 mg for adolescents 12 to 17 years of age at baseline in the preceding Core study NCT00619619.
Period: Overall Study
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Started | 20 | 20
Completed | 12 | 7
Not Completed | 8 | 13
Not completed — Adverse Event | 4 | 3
Not completed — Caregiver request | 3 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVS SR - Children | DVS SR - Adolescents | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.65 (1.31) | 13.55 (1.64) | 11.60 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 11 | 20
Number of participants for Tanner Assessment: Females [Number; unit: participants] — Female pubertal development of secondary sexual characteristics documented by pubic hair development and breast size (test categories). Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). N=9 Children, 9 Adolescent participants at observation. Participants may be represented in more than 1 test category.
  participants
    Breasts Stage 1 | 4 | 0 | 4
    Breasts Stage 2 | 4 | 1 | 5
    Breasts Stage 3 | 1 | 0 | 1
    Breasts Stage 4 | 0 | 1 | 1
    Breasts Stage 5 | 0 | 7 | 7
    Pubic hair Stage 1 | 6 | 0 | 6
    Pubic hair Stage 2 | 3 | 2 | 5
    Pubic hair Stage 3 | 0 | 0 | 0
    Pubic hair Stage 4 | 0 | 2 | 2
    Pubic hair Stage 5 | 0 | 5 | 5
Number of participants for Tanner Assessment: Males [Number; unit: participants] — Male pubertal development of secondary sexual characteristics documented by size of genitalia and pubic hair development (test categories). Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity, size). N=9 Children, 10 Adolescent participants at observation. Participants may be represented in > than 1 test category.
  participants
    Penis Stage 1 | 5 | 0 | 5
    Penis Stage 2 | 3 | 2 | 5
    Penis Stage 3 | 1 | 2 | 3
    Penis Stage 4 | 0 | 3 | 3
    Penis Stage 5 | 0 | 3 | 3
    Pubic hair Stage 1 | 6 | 0 | 6
    Pubic hair Stage 2 | 2 | 1 | 3
    Pubic hair Stage 3 | 1 | 3 | 4
    Pubic hair Stage 4 | 0 | 4 | 4
    Pubic hair Stage 5 | 0 | 2 | 2
    Testes Stage 1 | 5 | 0 | 5
    Testes Stage 2 | 2 | 1 | 3
    Testes Stage 3 | 2 | 3 | 5
    Testes Stage 4 | 0 | 3 | 3
    Testes Stage 5 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events AEs) and Serious Adverse Events (SAEs)
Description: AEs are any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study treatment. The event does not need to be causally related to the study treatment. SAEs are adverse events that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in persistent or significant disability or incapacity, result in cancer, or result in a congenital anomaly or birth defect.
Time Frame: Baseline (Extension study) up to Extension study Week 29 Follow up visit
Population: Safety population (Baseline=Extension study) includes all treatment assigned participants with at least 1 dose of study treatment during Extension study NCT00669110.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
participants
  Adverse events | 13 | 15
  Serious adverse events | 1 | 0

2. Primary Outcome: Number of Participants for Columbia Suicide-Severity Rating Scale (C-SSRS) According to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories
Description: C-SSRS is a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Yes/No responses are mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories: Completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. A participant could have a yes or no response in more than one category.
Time Frame: Postbaseline (≥Day 1 in Core study NCT00619619) up to Week 26 (Extension study)
Population: Safety population (Baseline=Core study) includes all treatment assigned participants with at least 1 dose of study treatment during Core study NCT00619619 and Extension study NCT00669110.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
participants
  Completed suicide: No | 20 | 20
  Suicide attempt: No | 20 | 20
  Preparatory acts - imminent suicidal behavior: No | 20 | 20
  Suicidal ideation: Yes | 0 | 3
  Suicidal ideation: No | 20 | 17
  Any suicidal behavior and/or ideation: Yes | 0 | 3
  Any suicidal behavior and/or ideation: No | 20 | 17
  Self-injurious behavior, no suicidal intent: No | 20 | 20

3. Other Pre Specified Outcome: Change From Baseline (Bsl) in Children's Depression Rating Scale - Revised (CDRS-R) Total Score at Final On-therapy Visit
Description: CDRS-R total score: scale measures 17 depressive symptoms, of which 3 are rated 1 to 5 and 14 are rated 1 to 7 (1 = no symptom difficulties; 5 to 7 = severe clinically significant difficulties) for a total score range of 17 to 113. Lower total scores indicate lower intensity of symptoms.
Time Frame: Baseline (Extension study), Extension study Outpatient Weeks 26 and >Week 26 (up to Week 29 or early termination)
Population: Intent to Treat population (ITT): all treatment assigned participants with a baseline primary efficacy evaluation, at least 1 dose of study treatment, and at least 1 primary efficacy evaluation after first dose in Extension study NCT00669110. Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
scores on a scale
  Baseline mean | 32.40 (7.61) | 33.70 (6.34)
  Change from Bsl Outpatient Week 26 | -1.85 (5.51) | -1.95 (6.85)
  Change from Bsl Outpatient Week >26 | -1.85 (5.51) | -1.70 (6.67)

4. Other Pre Specified Outcome: Percentage of Participants With Remission (Total Score ≤28) Based on Children's Depression Rating Scale - Revised (CDRS-R)
Description: CDRS-R total score: scale measures 17 depressive symptoms, of which 3 are rated 1 to 5 and 14 are rated 1 to 7 (1 = no symptom difficulties; 5 to 7 = severe clinically significant difficulties) for a total score range of 17 to 113. Lower total scores indicate lower intensity of symptoms. Remission defined as a CDRS-R total score ≤28 (coded value of 1).
Time Frame: Extension study Outpatient Weeks 1, 2, 4, 6, 10, 14, 18, 22, 26, and >26 (up to Week 29)
Population: ITT population; LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
percentage of participants
  Outpatient Week 1 | 26.7 | 21.1
  Outpatient Week 2 | 30 | 25
  Outpatient Week 4 | 30 | 20
  Outpatient Week 6 | 25 | 25
  Outpatient Week 10 | 45 | 25
  Outpatient Week 14 | 25 | 25
  Outpatient Week 18 | 35 | 40
  Outpatient Week 22 | 30 | 35
  Outpatient Week 26 | 30 | 30
  Outpatient Week >26 | 30 | 25

5. Other Pre Specified Outcome: Change From Baseline (Bsl) in Hamilton Rating Scale for Depression 17-item (HAM-D17) Total Score
Description: HAM-D17 is a clinician-rated interview to measure presence of depressive symptoms in 17 areas (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Total score ranges from 0 to 52; higher scores reflect higher severity of current illness states.
Time Frame: Baseline (Extension study), Extension study Outpatient Weeks 1, 2, 4, 6, 10, 14, 18, 22, 26, and >26 (up to Week 29)
Population: ITT population; LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
scores on a scale
  Baseline mean | 5.15 (3.01) | 7.45 (4.10)
  Change from Bsl Outpatient Week 1 | 0.53 (2.72) | 1.79 (2.97)
  Change from Bsl Outpatient Week 2 | -0.50 (2.80) | 0.70 (3.01)
  Change from Bsl Outpatient Week 4 | -0.40 (2.28) | -0.95 (2.24)
  Change from Bsl Outpatient Week 6 | -0.45 (2.31) | -0.70 (2.68)
  Change from Bsl Outpatient Week 10 | -1.30 (3.06) | -1.40 (2.66)
  Change from Bsl Outpatient Week 14 | -0.45 (2.58) | -1.65 (3.08)
  Change from Bsl Outpatient Week 18 | -1.65 (2.48) | -2.45 (3.10)
  Change from Bsl Outpatient Week 22 | -1.05 (2.26) | -2.15 (3.22)
  Change from Bsl Outpatient Week 26 | -1.65 (2.94) | -2.35 (3.39)
  Change from Bsl Outpatient Week >26 | -1.65 (2.94) | -2.10 (3.37)

6. Other Pre Specified Outcome: Percentage of Participants With a Categorical Clinical Global Impressions Scales - Severity (CGI-S) Score
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1=normal, not ill at all, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill patients. Higher scores reflect higher severity of current illness states.
Time Frame: Extension study Outpatient Weeks 1, 2, 4, 6, 10, 14, 18, 22, 26, and >26 (up to Week 29)
Population: ITT population; LOCF. No participants had a CGI-S score of 5, 6 or 7 (markedly, severely, or extremely ill), therefore only scores 1 through 4 (normal to moderately ill) are reported.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
percentage of participants
  Outpatient Week 1: not ill at all | 13.3 | 10.5
  Outpatient Week 1: borderline ill | 53.3 | 10.5
  Outpatient Week 1: mildly ill | 26.7 | 57.9
  Outpatient Week 1: moderately ill | 6.7 | 21.1
  Outpatient Week 2: not ill at all | 10 | 10
  Outpatient Week 2: borderline ill | 40 | 20
  Outpatient Week 2: mildly ill | 45 | 45
  Outpatient Week 2: moderately ill | 5 | 25
  Outpatient Week 4: not ill at all | 10 | 10
  Outpatient Week 4: borderline ill | 50 | 30
  Outpatient Week 4: mildly ill | 30 | 35
  Outpatient Week 4: moderately ill | 10 | 25
  Outpatient Week 6: not ill at all | 10 | 10
  Outpatient Week 6: borderline ill | 40 | 20
  Outpatient Week 6: mildly ill | 45 | 50
  Outpatient Week 6: moderately ill | 5 | 20
  Outpatient Week 10: not ill at all | 15 | 10
  Outpatient Week 10: borderline ill | 45 | 35
  Outpatient Week 10: mildly ill | 35 | 45
  Outpatient Week 10: moderately ill | 5 | 10
  Outpatient Week 14: not ill at all | 5 | 5
  Outpatient Week 14: borderline ill | 55 | 55
  Outpatient Week 14: mildly ill | 35 | 30
  Outpatient Week 14: moderately ill | 5 | 10
  Outpatient Week 18: not ill at all | 5 | 5
  Outpatient Week 18: borderline ill | 70 | 55
  Outpatient Week 18: mildly ill | 20 | 35
  Outpatient Week 18: moderately ill | 5 | 5
  Outpatient Week 22: not ill at all | 5 | 5
  Outpatient Week 22: borderline ill | 60 | 55
  Outpatient Week 22: mildly ill | 30 | 35
  Outpatient Week 22: moderately ill | 5 | 5
  Outpatient Week 26: not ill at all | 5 | 5
  Outpatient Week 26: borderline ill | 75 | 50
  Outpatient Week 26: mildly ill | 15 | 40
  Outpatient Week 26: moderately ill | 5 | 5
  Outpatient Week >26: not ill at all | 5 | 5
  Outpatient Week >26: borderline ill | 75 | 50
  Outpatient Week >26: mildly ill | 15 | 40
  Outpatient Week >26: moderately ill | 5 | 5

7. Other Pre Specified Outcome: Percentage of Participants With a Categorical Clinical Global Impressions Scales - Improvement (CGI-I) Score
Description: CGI-I: 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Scores above 4 reflect worsening of illness state as compared to baseline.
Time Frame: Baseline (Core study NCT00619619), Extension study Outpatient Weeks 1, 2, 4, 6, 10, 14, 18, 22, 26, and >26 (up to Week 29)
Population: ITT population; LOCF. No participants had a CGI-I score of 6 or 7 (much worse, very much worse), therefore only scores 1 through 5 (very much improved to minimally worse) are reported. CGI-I data for Inpatient Days 1 to 4 reported in Core study NCT00619619.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
percentage of participants
  Outpatient Week 1: very much improved | 25 | 10
  Outpatient Week 1: much improved | 55 | 45
  Outpatient Week 1: minimally improved | 20 | 40
  Outpatient Week 1: minimally worse | 0.0 | 5
  Outpatient Week 2: very much improved | 25 | 15
  Outpatient Week 2: much improved | 55 | 55
  Outpatient Week 2: minimally improved | 15 | 30
  Outpatient Week 4: very much improved | 35 | 20
  Outpatient Week 4: much improved | 45 | 55
  Outpatient Week 4: minimally improved | 15 | 25
  Outpatient Week 4: minimally worse | 5 | 0.0
  Outpatient Week 6: very much improved | 35 | 20
  Outpatient Week 6: much improved | 35 | 65
  Outpatient Week 6: minimally improved | 30 | 15
  Outpatient Week 10: very much improved | 30 | 30
  Outpatient Week 10: much improved | 40 | 50
  Outpatient Week 10: minimally improved | 30 | 15
  Outpatient Week 10: no change | 0.0 | 5
  Outpatient Week 14: very much improved | 25 | 40
  Outpatient Week 14: much improved | 50 | 40
  Outpatient Week 14: minimally improved | 20 | 15
  Outpatient Week 14: no change | 5 | 5
  Outpatient Week 18: very much improved | 30 | 40
  Outpatient Week 18: much improved | 55 | 45
  Outpatient Week 18: minimally improved | 15 | 15
  Outpatient Week 22: very much improved | 30 | 45
  Outpatient Week 22: much improved | 50 | 40
  Outpatient Week 22: minimally improved | 20 | 15
  Outpatient Week 26: very much improved | 40 | 40
  Outpatient Week 26: much improved | 45 | 45
  Outpatient Week 26: minimally improved | 15 | 15
  Outpatient Week >26: very much improved | 40 | 40
  Outpatient Week >26: much improved | 45 | 45
  Outpatient Week >26: minimally improved | 15 | 15

8. Other Pre Specified Outcome: Percentage of Participants With a Response of Much Improved or Very Much Improved Based on the Clinical Global Impressions Scales - Improvement (CGI-I) Score
Description: CGI-I: 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Participant with response is defined as having a score of 1 (very much improved) or 2 (much improved).
Time Frame: as for outcome 7
Population: ITT population; LOCF. CGI-I data for Inpatient Days 1 to 4 reported in Core study NCT00619619.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
percentage of participants
  Outpatient Week 1 | 80 | 55
  Outpatient Week 2 | 80 | 70
  Outpatient Week 4 | 80 | 75
  Outpatient Week 6 | 70 | 85
  Outpatient Week 10 | 70 | 80
  Outpatient Week 14 | 75 | 80
  Outpatient Week 18 | 85 | 85
  Outpatient Week 22 | 80 | 85
  Outpatient Week 26 | 85 | 85
  Outpatient Week >26 | 85 | 85

9. Other Pre Specified Outcome: Change From Baseline in Number of Participants for Tanner Assessment at Week 26: Females
Description: Tanner Children and Adolescent Pubertal Staging questionnaire used to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size (test categories). Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). Change categories: 0=no change in stage, 1=change of 1 stage, 2=change of 2 stages, 3=change of 3 stages, and 4=change of 4 stages. Participants may be represented in more than 1 test category.
Time Frame: Baseline (Extension study), Week 26 (Extension study)
Population: Safety population (Baseline=Extension study); N=number of participants with evaluable data at observation. No participants had a change of 3 stages or change of 4 stages reported, therefore only changes for 0 stages through 2 stages are reported.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 7 | 3
participants
  Breasts: 0=no stage change | 5 | 1
  Breasts: 1=change of 1 stage | 1 | 1
  Breasts: 2=change of 2 stages | 1 | 1
  Pubic hair: 0=no stage change | 6 | 2
  Pubic hair: 1=change of 1 stage | 1 | 0
  Pubic hair: 2=change of 2 stages | 0 | 1

10. Other Pre Specified Outcome: Change From Baseline in Number of Participants for Tanner Assessment at Week 26: Males
Description: Tanner Children and Adolescent Pubertal Staging questionnaire used to document the stage of development of secondary sexual characteristics. Male pubertal development staged by size of the genitalia and development of pubic hair (test categories). Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). Change categories: 0=no change in stage, 1=change of 1 stage, 2=change of 2 stages, 3=change of 3 stages, and 4=change of 4 stages. Participants may be represented in more than 1 test category.
Time Frame: Baseline (Extension study), Week 26 (Extension study)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 5 | 4
participants
  Penis: 0=no stage change | 4 | 3
  Penis: 1=change of 1 stage | 1 | 0
  Penis: 2=change of 2 stages | 0 | 1
  Pubic hair: 0=no stage change | 2 | 2
  Pubic hair: 1=change of 1 stage | 3 | 1
  Pubic hair: 2=change of 2 stages | 0 | 1
  Testes: 0=no stage change | 3 | 3
  Testes: 1=change of 1 stage | 2 | 0
  Testes: 2=change of 2 stages | 0 | 1

11. Other Pre Specified Outcome: Number of Participants With Vital Sign Results of Potential Clinical Importance (PCI): Blood Pressure (BP)
Description: PCI criteria for females: systolic BP [SBP] ranges from >110 and diastolic BP [DBP] >73 (>110/73) at age 6 up to BP >124/81 at age 11; BP from >121/79 at age 12 up to BP >132/86 at age 17. Criteria for males: BP ranges from >112/73 at age 6 up to BP >123/82 at age 10; BP from >119/79 at age 11 up to BP >140/89 at age 17. Vitals signs meeting the criteria for PCI categorized as BP elevation for 3 consecutive visits or as postural change in BP (decrease in SBP ≥20 millimeters of mercury [mmHg] or in DBP ≥15 mmHg for the last supine to first standing BP [supine to standing]).
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study).
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
participants
  Elevated supine SBP, 3 consecutive visits | 4 | 0
  Decrease SBP ≥20 mmHg supine to standing | 2 | 0
  Decrease DBP ≥15 mmHg supine to standing | 0 | 3

12. Other Pre Specified Outcome: Number of Participants With Vital Sign Results of Potential Clinical Importance (PCI): Weight
Description: Vitals signs meeting the PCI criteria for weight categorized according to an increase of ≥7 percent or a decrease of ≥3.5 percent in body weight.
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study).
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
participants
  Increase ≥7 percent in body weight | 11 | 4
  Decrease of ≥3.5 percent in body weight | 1 | 3

13. Other Pre Specified Outcome: Number of Participants With Vital Sign Results of Potential Clinical Importance (PCI): Pulse Rate
Description: PCI criteria for females: supine pulse rate (beats per minute [bpm]) ranges from <68 or >126 at age 6 to pulse <63 or >121 at age 11; pulse from <63 or >121 at age 12 to <54 or >110 at age 17; pulse from <50 or >104 at age 18. Criteria for males: pulse ranges from <68 or >126 at age 6 to pulse <63 or >121 at age 11; pulse from <58 or >116 at age 12 to <50 or >104 at age 17; pulse from <45 or >99 at age 18. Vitals signs meeting criteria for PCI categorized as Low or as postural change in pulse (increase in pulse ≥20 bpm for last supine to first standing pulse [supine to standing]).
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study).
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 20 | 20
participants
  Low supine pulse rate | 1 | 2
  Increase in pulse rate ≥20 mmHg supine to standing | 14 | 12

14. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Results of Potential Clinical Importance (PCI)
Description: ECG results meeting the criteria for PCI categorized as PR interval ≥200 milliseconds (msec); QT interval ≥480msec; QRS interval ≥120 msec; corrected QT (QTc) ≥500 msec ); >450 msec for males and >470 msec for females or increase of ≥60 msec or ≥30 msec change from baseline QTcB=QT corrected using Bazett formula; QTcF=QT corrected using the Fridericia formula.
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study). N=number of participants with analyzable ECG data. Participants may be represented in >1 category.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 17 | 14
participants
  PR interval ≥200 msec | 0 | 1
  QRS interval ≥120 msec | 0 | 1
  QTcF interval ≥30 msec change from baseline | 5 | 1
  QTcB interval ≥30 msec change from baseline | 6 | 1
  QTcB interval ≥60 msec change from baseline | 1 | 0
  QTcB interval >470 or increase ≥60 msec (females) | 1 | 0

15. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Results of Potential Clinical Importance (PCI): Heart Rate (Low)
Description: PCI criteria for females: heart rate (bpm) ranges from <68 and >126 at age 6 to <63 and >121 at age 11; heart rate from <63 and >121 at age 12 to <54 and >110 at age 17; heart rate <50 and >104 at age 18. Criteria for males: heart rate ranges from < 68 and >126 at age 6 to <63 and >121 at age 11; heart rate <58 and >116 at age 12 up <50 and >104 at age 17; heart rate <45 and >99 at age 18. Heart rates meeting the criteria for PCI categorized as low (less than the lower limit specified for age).
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study). N=number of participants with analyzable ECG data.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 17 | 14
participants | 0 | 2

16. Other Pre Specified Outcome: Number of Participants With Laboratory Test Results of Potential Clinical Importance (PCI)
Description: Laboratory test results meeting the criteria for PCI categorized as bicarbonate increase or decrease from baseline of ≥4 millimoles per liter (mmol/L); hematocrit <0.32 or >0.50 (females) or <0.37 or >0.55 (males) liters per liter (L/L); high density lipoprotein (HDL) cholesterol (fasting or nonfasting / unknown) decrease >0.21 mmol/L and test value ≥1.16 mmol/L; triglycerides (fasting or nonfasting / unknown) ≥2.258 mmol/L or increase ≥1.13 mmol/L and test value ≥3.39 mmol/L; urine specific gravity <1.001 or >1.035; and positive urinalysis result for protein (albumin), hemoglobin, or ketones.
Time Frame: Baseline (Extension study) up to Week 26 (Extension study)
Population: Safety population (Baseline=Extension study). N=number of participants with analyzable laboratory data. Participants may be represented in >1 category.
Measure: Number; unit: participants
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Number analyzed (Participants) | 17 | 14
participants
  Bicarbonate: increase | 2 | 0
  Bicarbonate: decrease | 0 | 1
  Hematocrit: low | 4 | 2
  HDL cholesterol: decrease | 2 | 1
  Triglycerides: high | 4 | 1
  Urine specific gravity: high | 3 | 3
  Urine protein albumin: positive result | 9 | 9
  Urine ketones: positive result | 0 | 1
  Urine hemoglobin: positive result | 0 | 1

ADVERSE EVENTS:
Time Frame: Events collected from the time of the signing of the informed consent form up to Week 29 (Follow up visit)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | DVS SR - Children | DVS SR - Adolescents
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR - Children (N=20) | DVS SR - Adolescents (N=20)
Negativism (oppositional behavior) (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | DVS SR - Children (N=20) | DVS SR - Adolescents (N=20)
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Feeling jittery (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Adenoiditis (Infections and infestations) | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastroenteritis viral infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Electrocardiogram abnormal (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 4 | 5
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 6
Syncope (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/11 | 1/9 — Female population
Aggression (Psychiatric disorders) | 2 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.